CLINICAL TRIAL: NCT05169814
Title: Micro/Nanobubbles (MNBs) and Wound Therapy: A Pilot Study Involving a Novel Oxygen Delivery System for Treatment of Acute and Chronic Wounds
Brief Title: Micro/Nanobubbles (MNBs) for Treatment of Acute and Chronic Wounds
Acronym: MNB
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Raj Vyas, Lead Investigator, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5901; 154138 (Other: FDA)
Record Dates: First submitted 2021-11-04; First posted 2021-12-27 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-06

CONDITIONS: Open Wound; Wound Heal
Keywords: acute wounds; chronic wounds; MNB solution; MNB; Micro/nanobubbles; Micronanobubbles; negative pressure wound therapy with instillation
MeSH Terms: interventions — Therapeutic Irrigation; Negative-Pressure Wound Therapy

STUDY DESIGN:
Intervention Model Description: This is a pilot study that consists of 4 arms:
  * Acute wounds: 1 control arm; 1 experimental arm (treated with MNB irrigation)
  * Chronic wounds: 1 control arm; 1 experimental arm (treated with Negative pressure wound therapy with MNB instillation)
Who Masked: Participant, Outcomes Assessor
Masking Description: This is a double-blind, controlled study. Participants will be selected and matched based on similar wound profiles, pathology mechanisms, comorbidity profiles, and age. They will randomly be assigned to the experimental (MNB) or control (normal saline) group. The randomization ratio between both groups will be 1:1. Measurements of objective datapoints (e.g. StO2), cytokines, proteases, and pH will be taken by blinded research personnel.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Acute Wounds - Control (Placebo Comparator): This arm will include patients with acute wounds and will receive standard of care: irrigation with normal saline.
  Interventions: Other: 0.9% Normal Saline - Irrigation
- Acute Wounds - Experimental (Experimental): This arm will include patients with acute wounds and will receive experimental treatment: irrigation with micro/nanobubbles (MNB's) in normal saline.
  Interventions: Drug: Micro/nanobubble (MNB) - Irrigation
- Chronic Wounds - Control (Placebo Comparator): This arm will include patients with chronic wounds and will receive standard of care: negative pressure wound therapy with instillation (NPWTi) using normal saline.
  Interventions: Other: 0.9% Normal Saline - Negative Pressure Wound Therapy with Instillation (NPWTi)
- Chronic Wounds - Experimental (Experimental): This arm will include patients with chronic wounds and will receive experimental treatment: negative pressure wound therapy with instillation (NPWTi) using micro/nanobubbles (MNB's) in normal saline.
  Interventions: Drug: Micro/nanobubble (MNB) - Negative Pressure Wound Therapy with Instillation (NPWTi)

INTERVENTIONS:
Drug: Micro/nanobubble (MNB) - Irrigation — An MNB solution will be used as an irrigation solution to improve wound oxygenation in ischemic tissue (e.g. ischemic surgical tissue, traumatic wounds, and failing replants). The MNB solution will be used in wet-to-dry wound care dressings with daily scheduled dressing changes.
  Arms: Acute Wounds - Experimental
Other: 0.9% Normal Saline - Irrigation — A normal saline solution will be used as an irrigation solution to improve wound oxygenation in ischemic tissue (e.g. ischemic surgical tissue, traumatic wounds, and failing replants). The normal saline solution will be used in wet-to-dry wound care dressings with daily scheduled dressing changes.
  Arms: Acute Wounds - Control
Drug: Micro/nanobubble (MNB) - Negative Pressure Wound Therapy with Instillation (NPWTi) — NPWTi with MNB will be applied to the wound with 20-minute instillation periods every 3 hours (standard instillation settings) with dressing changes every 3-5 days.
  Arms: Chronic Wounds - Experimental
Other: 0.9% Normal Saline - Negative Pressure Wound Therapy with Instillation (NPWTi) — NPWTi with normal saline will be applied to the wound with 20-minute instillation periods every 3 hours (standard instillation settings) with dressing changes every 3-5 days.
  Arms: Chronic Wounds - Control

SUMMARY:
The purpose of this study is to assess the safety and efficacy of Micro/nanobubbles (MNB's) for the healing of acute and chronic wounds.

DETAILED DESCRIPTION:
Oxygen delivery is one of the primary factors in wound healing. Micro/nanobubbles (MNBs) can be used to increase the oxygen dissolved in solution and increase oxygen delivery to a wound. The purpose of this research study is to determine if MNBs applied to a wound improve wound healing.

After being informed about the study and potential risks, all patients will need to provide written informed consent before being included in the study. The characteristics of the wound will be assessed and measurements will be taken before and after treatment. Depending on the patient's wound type, the patient will be treated with MNBs in saline gauze which will be applied to the wound daily (for acute wounds), or MNBs in negative pressure wound therapy with instillation (NPWTi) (for chronic wounds) which will be applied to the wound continuously throughout the day with the wound evaluated and sponge replaced every 3-5 days. This is consistent with the current standard of wound care with gauze or NPWTi. Tissue oxygenation using infrared technology and wound healing will be measured and results collected for analysis.

Participation will last approximately 2-4 weeks or the duration of the inpatient admission. If discharge from the hospital is earlier than 2 weeks, the treatment will be discontinued and results will be submitted for analysis.

ELIGIBILITY:
Inclusion Criteria:

* are above the age of 18.
* have traumatic, surgical, or chronic wounds.
* have radiotherapy related tissue injury.
* have thermal, chemical, and/or electrical burn injuries.
* have pressure ulcers, diabetic foot ulcers, venous ulcers, arterial ulcers, and/or neuropathic skin ulcers.
* have acute ischemic wounds

Exclusion Criteria:

* have infected wounds.
* have wounds with exposed vital structures such as nerves, arteries, and/or veins.
* have wounds associated with malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-10-09 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Wound total oxygen saturation level | 2-4 weeks
  Near Infrared Spectroscopy Imaging (NIRS) (KENT SnapShot https://www.kentimaging.com/product/) will be used to assess wound oxygenation saturation levels prior to the MNB or normal saline application. This will provide the investigators with a baseline oxygen saturation measurement. The NIRS KENT SnapShot is an FDA approved non-contact-based imaging modality used to assess wound/tissue oxygenation in the clinical setting and is currently available in the investigators' research laboratory.
Wound Size/ Surface Area (cm^2) | 2-4 weeks
  Daily photographs taken before initiation of treatment and during treatment.
Analysis of wound pH | 2-4 weeks
  With each dressing change, a non-traumatic vidal curette will be used to collect wound exudate in both groups, and a pH strip will be used to measure the pH.
Wound oxyhemoglobin concentration level | 2-4 weeks
  Near Infrared Spectroscopy Imaging (NIRS) (KENT SnapShot https://www.kentimaging.com/product/) will be used to assess wound oxyhemoglobin concentration levels prior to the MNB or normal saline application. This will provide the investigators with a baseline oxygen tension measurement. The NIRS KENT SnapShot is an FDA approved non-contact-based imaging modality used to assess wound/tissue oxygenation in the clinical setting and is currently available in the investigators' research laboratory.
Wound deoxyhemoglobin concentration level | 2-4 weeks
  Near Infrared Spectroscopy Imaging (NIRS) (KENT SnapShot https://www.kentimaging.com/product/) will be used to assess wound deoxyhemoglobin concentration levels prior to the MNB or normal saline application. This will provide the investigators with a baseline oxygen tension measurement. The NIRS KENT SnapShot is an FDA approved non-contact-based imaging modality used to assess wound/tissue oxygenation in the clinical setting and is currently available in the investigators' research laboratory.
Analysis of wound GM-CSF concentration level | 2-4 weeks
  With each dressing change, a non-traumatic vidal curette will be used to collect wound exudate in both groups. The proteins will then be extracted by standard methods, and ELISA kits will be used to assess GM-CSF concentration levels.
Analysis of wound interferon concentration levels | 2-4 weeks
  With each dressing change, a non-traumatic vidal curette will be used to collect wound exudate in both groups. The proteins will then be extracted by standard methods, and ELISA kits will be used to assess the following interferon concentration levels: IFN alpha, IFN gamma.
  *These levels will be reported in the same units of measure.
Analysis of wound interleukin (IL) concentration levels | 2-4 weeks
  With each dressing change, a non-traumatic vidal curette will be used to collect wound exudate in both groups. The proteins will then be extracted by standard methods, and ELISA kits will be used to assess the following interleukin concentration levels: IL-1 alpha, IL-1 beta, IL-1RA, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8 (CXCL8), IL-9, IL-10, IL-12p70, IL-13, IL-15, IL-17A (CTLA-8), IL-18, IL-21, IL-22, IL-23, IL-27, IL-31.
  *These levels will be reported in the same units of measure.
Analysis of wound tumor necrosis factor (TNF) concentration levels | 2-4 weeks
  With each dressing change, a non-traumatic vidal curette will be used to collect wound exudate in both groups. The proteins will then be extracted by standard methods, and ELISA kits will be used to assess the following TNF concentration levels: TNF alpha, TNF beta.
  *These levels will be reported in the same units of measure.
Analysis of wound Eotaxin (CCL11) concentration level | 2-4 weeks
  With each dressing change, a non-traumatic vidal curette will be used to collect wound exudate in both groups. The proteins will then be extracted by standard methods, and ELISA kits will be used to assess Eotaxin (CCL11) concentration levels.
Analysis of wound GRO alpha (CXCL1) concentration level | 2-4 weeks
  With each dressing change, a non-traumatic vidal curette will be used to collect wound exudate in both groups. The proteins will then be extracted by standard methods, and ELISA kits will be used to assess GRO alpha (CXCL1) concentration levels.
Analysis of wound IP-10 (CXCL10) concentration level | 2-4 weeks
  With each dressing change, a non-traumatic vidal curette will be used to collect wound exudate in both groups. The proteins will then be extracted by standard methods, and ELISA kits will be used to assess IP-10 (CXCL10) concentration levels.
Analysis of wound MCP-1 (CCL2) concentration level | 2-4 weeks
  With each dressing change, a non-traumatic vidal curette will be used to collect wound exudate in both groups. The proteins will then be extracted by standard methods, and ELISA kits will be used to assess MCP-1 (CCL2) concentration levels.
Analysis of wound MIP-1 alpha (CCL3) concentration level | 2-4 weeks
  With each dressing change, a non-traumatic vidal curette will be used to collect wound exudate in both groups. The proteins will then be extracted by standard methods, and ELISA kits will be used to assess MIP-1 alpha (CCL3) concentration levels.
Analysis of wound MIP-1 beta (CCL4) concentration level | 2-4 weeks
  With each dressing change, a non-traumatic vidal curette will be used to collect wound exudate in both groups. The proteins will then be extracted by standard methods, and ELISA kits will be used to assess MIP-1 beta (CCL4) concentration levels.
Analysis of wound RANTES (CCL5) concentration level | 2-4 weeks
  With each dressing change, a non-traumatic vidal curette will be used to collect wound exudate in both groups. The proteins will then be extracted by standard methods, and ELISA kits will be used to assess RANTES (CCL5) concentration levels.
Analysis of wound SDF-1 alpha concentration level | 2-4 weeks
  With each dressing change, a non-traumatic vidal curette will be used to collect wound exudate in both groups. The proteins will then be extracted by standard methods, and ELISA kits will be used to assess SDF-1 alpha concentration levels.
Analysis of wound matrix metalloproteinase 1 (MMP1) concentration level | 2-4 weeks
  With each dressing change, a non-traumatic vidal curette will be used to collect wound exudate in both groups. The proteins will then be extracted by standard methods, and ELISA kits will be used to assess MMP1 concentration level.
Analysis of wound matrix metalloproteinase 8 (MMP8) concentration level | 2-4 weeks
  With each dressing change, a non-traumatic vidal curette will be used to collect wound exudate in both groups. The proteins will then be extracted by standard methods, and ELISA kits will be used to assess MMP8 concentration level.
Analysis of wound matrix metalloproteinase 13 (MMP13) concentration level | 2-4 weeks
  With each dressing change, a non-traumatic vidal curette will be used to collect wound exudate in both groups. The proteins will then be extracted by standard methods, and ELISA kits will be used to assess MMP 13 concentration level.

SECONDARY OUTCOMES:
Hospital Length of Stay (LOS) | 2-4 weeks
  Days of hospital admission
Number of participants that return to the operating room | 2-4 weeks
  Qualifying individuals include participants that return to the operating room for a procedure (e.g. surgical debridement) on the same wound being treated by the study investigators.
Number of participants readmitted to the hospital for same wound after discharge | 4-8 weeks
  Qualifying individuals include participants that are readmitted to the hospital for the same wound that was treated by the study investigators.

CONTACTS AND LOCATIONS:
Overall Officials: Raj Vyas, MD, Principal Investigator — University of California, Irvine, Dept. of Plastic Surgery; Vice-Chairman
Locations (1):
- UCI Medical Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers outside this study.

REFERENCES:
- [Background] Tsuge H. Micro- and Nanobubbles: Fundamentals and Applications. Boca Raton: CRC Press; 2014.
- [Background] Matiasek J, Djedovic G, Kiehlmann M, Verstappen R, Rieger UM. Negative pressure wound therapy with instillation: effects on healing of category 4 pressure ulcers. Plastic and Aesthetic Research. 2018;5.
- [Result] Sayadi LR, Banyard DA, Ziegler ME, Obagi Z, Prussak J, Klopfer MJ, Evans GR, Widgerow AD. Topical oxygen therapy & micro/nanobubbles: a new modality for tissue oxygen delivery. Int Wound J. 2018 Jun;15(3):363-374. doi: 10.1111/iwj.12873. Epub 2018 Jan 5. PMID 29314626
- [Result] Khan MS, Hwang J, Lee K, Choi Y, Kim K, Koo HJ, Hong JW, Choi J. Oxygen-Carrying Micro/Nanobubbles: Composition, Synthesis Techniques and Potential Prospects in Photo-Triggered Theranostics. Molecules. 2018 Aug 31;23(9):2210. doi: 10.3390/molecules23092210. PMID 30200336
- [Result] Lalezari S, Lee CJ, Borovikova AA, Banyard DA, Paydar KZ, Wirth GA, Widgerow AD. Deconstructing negative pressure wound therapy. Int Wound J. 2017 Aug;14(4):649-657. doi: 10.1111/iwj.12658. Epub 2016 Sep 29. PMID 27681204
- [Result] Back DA, Scheuermann-Poley C, Willy C. Recommendations on negative pressure wound therapy with instillation and antimicrobial solutions - when, where and how to use: what does the evidence show? Int Wound J. 2013 Dec;10 Suppl 1(Suppl 1):32-42. doi: 10.1111/iwj.12183. PMID 24251842
- [Result] Jarbrink K, Ni G, Sonnergren H, Schmidtchen A, Pang C, Bajpai R, Car J. The humanistic and economic burden of chronic wounds: a protocol for a systematic review. Syst Rev. 2017 Jan 24;6(1):15. doi: 10.1186/s13643-016-0400-8. PMID 28118847

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-08): https://cdn.clinicaltrials.gov/large-docs/14/NCT05169814/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-08): https://cdn.clinicaltrials.gov/large-docs/14/NCT05169814/ICF_001.pdf